CLINICAL TRIAL: NCT06020339
Title: The Effect of the Education Given to Primiparous Pregnant Women Within the Framework of the Continuous Midwifery Care Model on Their Fears of Birth, Birth Preferences and Postpartum Trauma Perceptions.
Brief Title: The Effect of the Continuous Midwifery Care Model on Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Özlem KOÇ, Educational Institution, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: suleozlem2023
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2023-11

CONDITIONS: Birth, First; Pregnancy Related; Newborn; Fit; Trauma, Psychological; Birth Trauma
Keywords: birth; midwifery care model; birth trauma; post traumatic stress disorder; pregnancy education
MeSH Terms: conditions — Psychological Trauma; Birth Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled longitudinal study. Within the framework of the prenatal continuous midwifery care model, pregnant women who will participate in four modules of training will form the study (education) group and those who do not will form the control group.
Who Masked: Participant
Masking Description: The sample of the study will consist of 80 pregnant women (40 Study Group: trained, 40 Control Group: not trained), who applied to the hospital between the dates of the study, who met the inclusion criteria and accepted to participate voluntarily in the study. The sample of the first 40 pregnant women to be included in the study (20 study-20 control) will be formed in the first 1st and 3rd month of the research, and the creation of the second sample of 40 pregnant women (20 study-20 control) will be done in the 12th and 13th months of the research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Randomization group (Experimental): Pregnant women in the study group will be given a total of 4 modules, 3 modules during pregnancy and 1 module in the postpartum period;
  * 1. module 20-28. During pregnancy weeks, trainings are in the form of face-to-face group training,
  * 2. module 29-36. During pregnancy weeks, trainings are in the form of face-to-face group training,
  * 3. module trainings 37-40. in the form of video-conference (zoom meeting) during pregnancy weeks,
  * 4. module will be applied in 1 month postpartum with face-to-face interview technique).
  Pregnancy 20-28. Pregnant women between weeks 29-36 should attend the 1st module education. 2nd module training in gestational weeks, 37-40. They will be trained in the 3rd module during the pregnancy weeks.
  module training will be individualized during the mother's visit in the 1st month postpartum.
  Version B (WDEQ) will be administered after the program is completed, and the Birth-Related Trauma Perception Scale will be administered after birth.
  Interventions: Other: The midwife-led continuous care model (MLCC)
- Control group (No Intervention): Pregnant women who will be included in the control group will receive routine midwifery care. In the postpartum period (WDEQ), version B and the Birth Trauma Perception Scale will be used.
  The pregnant women will inform the researcher by telephone after the birth (within the first 24 hours) and the mother will be visited by the researcher within the first month after the birth, and the trauma perceptions of the mothers will be evaluated with the Birth Trauma Perception Scale.

INTERVENTIONS:
Other: The midwife-led continuous care model (MLCC) — Continuity of midwife-led care has been defined as care in which the midwife is the leading professional in the planning, organization and delivery of care given to a woman from the initial assessment of the pregnant woman to the postpartum period.
  ELSBM; It is the same midwife or midwife group providing the care and counseling needed by the woman during pregnancy, childbirth and postpartum period. In this care model, the midwife is the leading health care specialist who is responsible for planning and arranging the care given to women in the antenatal, natal and postnatal period. MLCC is woman-centered and is based on the idea that pregnancy and childbirth are normal life events.
  This care model includes education, counseling and care according to the needs of the woman. It promotes vaginal delivery as a normal process and advocates minimal interventions. Continuity of midwifery-led care is associated with superior outcomes for women and infants than other models of care.
  Other Names: Midwife-Led Care
  Arms: Randomization group

SUMMARY:
It is the right of both the mother and her baby to receive the best care and give birth in the best way possible for every pregnant woman. World Health Organization midwife; It defines a person trained to provide necessary care and counseling during pregnancy, at birth and after birth, to have normal births under his own responsibility, to care for the newborn and to provide family planning counseling. According to the Ministry of Health, the midwife provides these services as well as immunization, protection from infectious and social diseases, etc. He is a healthcare professional who fulfills his roles.

However, in our country, pregnancy, birth and postpartum care services are primarily carried out under the control of a physician, and most of them include medical follow-up. The routine care given by midwives to pregnant women during pregnancy is unfortunately limited to performing the procedures and cannot adequately meet the needs of the woman. As a result, cesarean section rates in our country have risen well above the acceptable level by WHO. Studies have shown that the rate of cesarean section increases with the number of pregnant women who apply to the doctor for pregnancy control. Turkey is the country with the highest cesarean section rates among OECD countries. According to the 2018 results of the Turkey Demographic and Health Survey (TNSA), the rate of cesarean section in our country is 52%. The World Health Organization (WHO) recommended 10-15% cesarean section rate in terms of maternal and infant health in 1985, and re-evaluated this recommendation in 2015. Women who have had a cesarean delivery have greater risks compared to women who have had a vaginal delivery. One of the most common complications after cesarean section is sepsis, and maternal mortality rates increase due to complications such as bleeding and infection after cesarean section. In addition, the choice of cesarean section, which negatively affects many variables such as epigenetically transmitted fear of birth and traumatic birth perception, breastfeeding and microbiota of the baby, is an important factor that will affect future generations. Cesarean section rates, which also cause high maternal and neonatal complication rates, have become a problem that increases health expenditures economically all over the world.

However, cesarean section rates are decreasing in countries where midwives play an active role in pregnancy follow-up. In the midwife-led continuous care model (MLCC), which is carried out by midwives, especially in countries with high normal birth rates, care is completely woman-centered. The model advocates vaginal delivery, which is the most superior form of delivery for maternal and infant health. Studies show that midwife-led continuous care increases vaginal birth rates, women experience a more positive birth, and reduces many unnecessary medical interventions. Within the scope of this care model, midwives train pregnant women from the beginning of pregnancy to the postpartum period and minimize their fear of childbirth based on the fear of the unknown. Another advantage of MLCC is that care will be given by the same midwife or midwife group. This ensures a good bond and uninterrupted communication between the woman and her midwife. This maintenance model is not yet used in our country. The study to be carried out with this training process planned within the scope of MLCC is unique in that it will be carried out for the first time at the national level.

The aim of the study is to evaluate the effect of training to be given with MLCC in reducing cesarean section preferences.

DETAILED DESCRIPTION:
The project has a unique value for a sustainable future in terms of the fear of birth, birth preference, birth perceptions of pregnant women in particular, and its effects at the social level in general. Another unique value is that it is a longitudinal study that uses innovative methods to be taken at the national level to quickly compensate for the acceleration lost in normal birth rates, especially during the pandemic process.

If this research is completed successfully, the researcher will have broken a new ground nationally. This success will contribute to the academic career and prestige of the researcher. The researcher plans to carry out ELSBM trainings, which she plans to start with a motto that supports vaginal birth, in special groups such as immigrant women, women with risky pregnancies, and in cooperation with different institutions in wider masses. As a result of the research, pregnant women participating in the research will receive qualified pregnancy and postpartum care. It is thought that this situation will increase the satisfaction of pregnant women with the institution and increase their preference for vaginal delivery. Thus, it is thought that it will contribute to the reduction of cesarean delivery rates, which have become a worldwide problem, cause high maternal and neonatal complication rates, and increase health expenditures economically.

The study was planned to be conducted with 80 pregnant women (experimental group 40-control group 40) in a randomized controlled manner. G*Power analysis was used to determine the sample size. In this study, it is planned to provide 4 modules of training to primiparous pregnant women within the framework of the midwife-led continuous care model (MLCC). The first 2 modules of the training to be given in the research were planned to be face-to-face training, the 3rd module as video-conference, and the 4th module as face-to-face training in the postpartum period.

If MLCC is integrated into the health care system, every mother will receive the quality care and education she deserves. This situation will reduce the fear of childbirth experienced by women and the perception of traumatic birth, and will direct women to vaginal birth. Vaginal delivery, which is superior in terms of both maternal and newborn health, has a lower cost compared to cesarean section. Thus, it is thought that MLCC, which will be a cost-effective care model within the scope of health services, will also benefit the country's economy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who have completed at least primary education,
* Able to speak, understand and write Turkish,
* Pregnant women between the ages of 18-35 (pregnant women under 18 and over 35 years of age will not be preferred since they are among the risky groups in terms of maternal and fetal)
* Pregnant women residing within the borders of Mersin-Tarsus
* Primigravidas (It is planned to include primigravidas in the study, considering that there may be different variables affecting the fear of childbirth in previous pregnancies of multiparas.)
* Pregnant women who do not have any obstacles to give vaginal birth
* Pregnant women with a single and healthy fetus will be included in the study.

Exclusion Criteria:

* Pregnant women with any risky pregnancy history (preeclampsia, placenta previa, gestational diabetes mellitus, oligohydramnios and polyhydramnios, etc.),
* Pregnant women with systemic and/or neurological disease,
* Pregnant women with cesarean indication,
* Pregnant women with chronic and/or psychiatric health problems (based on self-report and clinical diagnosis),
* Pregnant women who participated in any childbirth preparation training program

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | through study completion, an average of 1 year
  It consists of questions about the sociodemographic characteristics, pregnancy and birth characteristics of the pregnant women who were prepared by the researcher by scanning the relevant literature.
VIJMA Birth expectation/experience Scale Version A | through study completion, an average of 1 year
  In order to determine the fear of childbirth, Wij-ma et al. (1998) developed by. The validity and reliability study of the scale in Turkish was performed by Korukcu et al. (2012) by It is an item scale. The scale has certain breakpoints. These; low-grade fear of childbirth (≤37), moderate-grade fear of childbirth (38-65), severe fear of childbirth (66-84), and clinical-grade fear of childbirth (≥85). In the validity-reliability study of the scale, the Cronbach Alpha value was found to be 0.89.

SECONDARY OUTCOMES:
Wijma Birth Expectation/Experience Scale B Version (Appendix-3) | through study completion, an average of 1 year
  The Turkish adaptation of the scale, which was first developed by K. Wijma et al. (2002), was made by Uçar and Beji in 2013. The scale includes fear, confidence, feeling of loneliness, happiness, etc. It consists of 33 questions in total, including feelings and thoughts. Each item is in a 6-point Likert type, scoring between 1 and 6. 1 is expressed as "totally" and 6 as "not at all". While the minimum-candle score is 33 on the scale, the maximum score is 198. High scores indicate that women's fear of childbirth is high. Negatively charged items (2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27, 31) in the scale are calculated by inverting them in order to ensure consistency in the measurement. In the study conducted by Wijma et al. (1998), Cronbach's alpha values were determined as 0.89 in nulliparas, 0.99 in multiparas and 0.93 in total. In the Turkish version, the Cronbach alpha value of the Wijma Birth Expectation/Experience Scale Version B was found to be 0.88.
Birth-Related Trauma Perception Scale | through study completion, an average of 1 year
  The Birth Trauma Perception Scale was developed by Mucuk and Ozkan to evaluate mothers' perceptions of trauma associated with vaginal delivery and can be used throughout the country as a valid and reliable measurement tool. The Birth Trauma Perception Scale can be used from the first postpartum week to one year. It is thought that the scale will enable the identification of individuals sensitive to trauma associated with birth, their evaluation in terms of trauma symptoms in the process, and the better quality of individualized midwifery care required in this regard. The scale is in a five-point Likert model. Total scale scores vary between 39-195. An increase in the score obtained from the scale indicates that the woman's perception of trauma is high. In the validity-reliability study of the scale, the Cronbach Alpha value was found to be 0.92.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem KOÇ, Study Chair — Tarsus University
Locations (1):
- Tarsus University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No